CLINICAL TRIAL: NCT01861821
Title: Prospective, Controlled, Randomized, Blinded, Single-center Study of the Clinical Efficacy and Outcomes of a Multiport Versus Uniport Flexible Catheter for Epidural Analgesia During Labor and Delivery
Brief Title: Analgesic Efficacy of a Multiport Versus Uniport Flexible Catheter for Labor Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 010-158
Record Dates: First submitted 2012-06-01; First posted 2013-05-24 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2016-09

CONDITIONS: Labor Pain
Keywords: Epidural catheter; Epidural analgesia; Labor epidural analgesia; Analgesic efficacy; Multiport epidural catheter; Uniport epidural catheter; Flexible epidural catheter
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Multiport flexible catheter (Active Comparator): Multiport flexible catheter has three ports for the delivery of epidural medication for labor analgesia
  Interventions: Device: Multiport flexible catheter
- Uniport flexible catheter (Active Comparator): Uniport flexible catheter has one port for the delivery of epidural medication for labor analgesia
  Interventions: Device: Uniport flexible catheter

INTERVENTIONS:
Device: Multiport flexible catheter — Multiport flexible catheter has three ports for the delivery of epidural medication
  Arms: Multiport flexible catheter
Device: Uniport flexible catheter — Uniport flexible catheter has one port for the delivery of epidural medication
  Arms: Uniport flexible catheter

SUMMARY:
The purpose of this study is to determine whether multiple ports improve the analgesic efficacy of flexible catheters used for the provision of epidural analgesia during the entire continuum of labor and delivery

DETAILED DESCRIPTION:
Multiport catheters, when compared to uniport catheters, have been associated with better analgesic quality during labor epidural analgesia because the presence of more than one port may enhance the distribution of epidural medication

Flexible catheters, when compared to rigid catheters, have been associated with better analgesic quality during labor epidural analgesia because greater flexibility may minimize catheter deviation in the epidural space, facilitate more optimal catheter placement in the epidural space, and result in better distribution of epidural medication

It is unknown whether multiple ports, which promote better distribution of epidural medication, provide added analgesic benefit to flexible catheters, which also facilitate better distribution of epidural medication, when used for the provision of epidural analgesia during labor and delivery

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification I-III parturients
* Mixed parity
* Estimated gestational age of at least 37 weeks
* Singleton gestation
* Cephalic presentation
* Spontaneous or induced labor

Exclusion Criteria:

* Body mass index (BMI) > 45 kg/m2
* Prior cesarean section
* Multiple gestation
* Fetal abnormality
* Use of chronic analgesic medication
* Local anesthetic allergy
* Coagulopathy or anticoagulation
* Infection at epidural insertion site
* Spinal deformity other than mild scoliosis
* Uncontrolled/uncompensated/uncorrected cerebral, cardiovascular, pulmonary, gastrointestinal, hepatic, renal, endocrinologic, metabolic, or hematologic condition

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 650 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Analgesic success rate | 30 minutes following the initiation of labor epidural analgesia
  Complete analgesia is defined as the complete relief of pain during contractions following the administration of the above epidural medication without requiring further epidural medication/intervention.

SECONDARY OUTCOMES:
Number of Clinician interventions during the first stage of labor | The duration of first stage of labor, an expected average of 6 hours and 30 minutes
  Clinician administered rescue epidural boluses during first stage of labor
Anesthetic success rate | 10 minutes following the initiation of epidural anesthesia for cesarean delivery
  Incidence of adequate anesthesia at initiation of epidural anesthesia for cesarean delivery
Maternal satisfaction with the overall quality of analgesia/anesthesia during labor and delivery | 24 hours following delivery
  Subjects will be asked to evaluate the quality of labor and delivery analgesia/anesthesia as: Poor, Fair, Good, Very good, Excellent

CONTACTS AND LOCATIONS:
Overall Officials: John Philip, MD, Principal Investigator — Baylor Scott and White Health
Locations (1):
- Baylor All Saints Medical Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Angelo R, Foss ML, Livesay CH. A comparison of multiport and uniport epidural catheters in laboring patients. Anesth Analg. 1997 Jun;84(6):1276-9. doi: 10.1097/00000539-199706000-00019. PMID 9174306
- [Background] Segal S, Eappen S, Datta S. Superiority of multi-orifice over single-orifice epidural catheters for labor analgesia and cesarean delivery. J Clin Anesth. 1997 Mar;9(2):109-12. doi: 10.1016/S0952-8180(97)00232-8. PMID 9075034
- [Background] Collier CB, Gatt SP. Epidural catheters for obstetrics. Terminal hole or lateral eyes? Reg Anesth. 1994 Nov-Dec;19(6):378-85. PMID 7848946
- [Background] Michael S, Richmond MN, Birks RJ. A comparison between open-end (single hole) and closed-end (three lateral holes) epidural catheters. Complications and quality of sensory blockade. Anaesthesia. 1989 Jul;44(7):578-80. doi: 10.1111/j.1365-2044.1989.tb11446.x. PMID 2774123
- [Background] Jaime F, Mandell GL, Vallejo MC, Ramanathan S. Uniport soft-tip, open-ended catheters versus multiport firm-tipped close-ended catheters for epidural labor analgesia: a quality assurance study. J Clin Anesth. 2000 Mar;12(2):89-93. doi: 10.1016/s0952-8180(00)00116-1. PMID 10818320
- [Background] Banwell BR, Morley-Forster P, Krause R. Decreased incidence of complications in parturients with the arrow (FlexTip Plus) epidural catheter. Can J Anaesth. 1998 Apr;45(4):370-2. doi: 10.1007/BF03012031. PMID 9597214
- [Background] Spiegel JE, Vasudevan A, Li Y, Hess PE. A randomized prospective study comparing two flexible epidural catheters for labour analgesia. Br J Anaesth. 2009 Sep;103(3):400-5. doi: 10.1093/bja/aep174. Epub 2009 Jun 27. PMID 19561345
- [Background] Hardy PA. Force exerted by epidural catheters. Anaesthesia. 1986 Mar;41(3):306-8. doi: 10.1111/j.1365-2044.1986.tb12794.x. PMID 3963335
- [Background] Hogan Q. Epidural catheter tip position and distribution of injectate evaluated by computed tomography. Anesthesiology. 1999 Apr;90(4):964-70. doi: 10.1097/00000542-199904000-00006. PMID 10201664
- [Background] McAtamney D, O'Hare C, Fee JP. An in vitro evaluation of flow from multihole epidural catheters during continuous infusion with four different infusion pumps. Anaesthesia. 1999 Jul;54(7):664-9. doi: 10.1046/j.1365-2044.1999.00892.x. PMID 10417459
- [Background] Chiron B, de Serres TM, Fusciardi J, Laffon M. Difficult Removal of an Arrow FlexTip Plus epidural catheter. Anesth Analg. 2008 Sep;107(3):1085-6. doi: 10.1213/ane.0b013e31817e038b. No abstract available. PMID 18713938
- [Background] Asai T, Shingu K. Advantages and disadvantages of the Arrow FlexTip Plus epidural catheter. Anaesthesia. 2001 Jun;56(6):606. No abstract available. PMID 11412201
- [Background] Hopf B, Leischik M. More on problems with removing the arrow FlexTip epidural catheter: smooth in-hardly out? Anesthesiology. 2000 Nov;93(5):1362. doi: 10.1097/00000542-200011000-00037. No abstract available. PMID 11046232
- [Background] Asai T, Sakai T, Murao K, Kojima K, Shingu K. More difficulty in removing an arrow epidural catheter. Anesth Analg. 2006 May;102(5):1595-6. doi: 10.1213/01.ANE.0000215172.96873.43. No abstract available. PMID 16632862
- [Background] Asai T, Yamamoto K, Hirose T, Taguchi H, Shingu K. Breakage of epidural catheters: a comparison of an arrow reinforced catheter and other nonreinforced catheters. Anesth Analg. 2001 Jan;92(1):246-8. doi: 10.1097/00000539-200101000-00048. No abstract available. PMID 11133637
- [Background] Bastien JL, McCarroll MG, Everett LL. Uncoiling of Arrow Flextip plus epidural catheter reinforcing wire during catheter removal: an unusual complication. Anesth Analg. 2004 Feb;98(2):554-555. doi: 10.1213/01.ANE.0000077718.21575.F6. No abstract available. PMID 14742413
- [Background] Pierre HL, Block BM, Wu CL. Difficult removal of a wire-reinforced epidural catheter. J Clin Anesth. 2003 Mar;15(2):140-1. doi: 10.1016/s0952-8180(02)00516-0. PMID 12719055
- [Background] Woehlck HJ, Bolla B. Uncoiling of wire in arrow flextip epidural catheter on removal. Anesthesiology. 2000 Mar;92(3):907-9. doi: 10.1097/00000542-200003000-00058. No abstract available. PMID 10719987